CLINICAL TRIAL: NCT00641290
Title: Cardiac Output and Central Venous Oxygen Saturation Monitoring Using the Vigileo FloTrac Sensor Versus Conventional Thermodilution Method Using the Pulmonary Artery Catheter: A Prospective Study
Brief Title: Vigileo FloTrac vs Pulmonary Artery Catheter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Sultanah Aminah Johor Bahru (Other Government)
Responsible Party: Dr. Gunalan Palari Arumugam, Hospital Sultanah Aminah Johor Bahru
Other Study IDs: NMRR ID 08-645-1800
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Ischemic Heart Disease; Valvular Heart Disease
Keywords: CABG; Valve surgery
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Vigileo FloTrac Sensor — Comparing the Vigileo FloTrac against the conventional Pulmonary Artery Catheter using the thermodilution method for measurements of cardiac output.

SUMMARY:
To study the role of Vigileo monitor using the FloTrac sensor to measure cardiac output using the pulse contour analysis as well as central venous oxygen saturation monitoring as a guide for tissue perfusion. The accuracy of the Vigileo monitoring was compared with the conventional thermodilution method for measuring cardiac output using the pulmonary artery catheter and mixed venous oxygen saturation for assessing global tissue perfusion.

DETAILED DESCRIPTION:
Cardiac Output and Central Venous Oxygen Saturation Monitoring Using the Vigileo FloTrac Sensor Versus Conventional Thermodilution Method Using the Pulmonary Artery Catheter: A Prospective Study

OBJECTIVE: To study the role of Vigileo monitor using the FloTrac sensor to measure cardiac output using the pulse contour analysis as well as central venous oxygen saturation monitoring as a guide for tissue perfusion. The accuracy of the Vigileo monitoring was compared with the conventional thermodilution method for measuring cardiac output using the pulmonary artery catheter and mixed venous oxygen saturation for assessing global tissue perfusion.

DESIGN: A prospective clinical study conducted at the cardiothoracic operating theatre and the cardiothoracic intensive care unit of Sultanah Aminah Hospital Johor Bahru.

PARTICIPANTS: 60 patients from the time of induction of anaesthesia to post operative Day 1 in the cardiothoracic intensive care unit.

INTERVENTIONS: Simultaneous cardiac output measurements using the Vigileo FloTrac sensor and thermodilution method using the PAC will be obtained at the following intervals: Post Induction( T0), Pre CPB( T1), Post CPB( T2), 1 hour post ICU admission( T3), 4 hours post ICU admission( T4), 1 hour post extubation( T5) and post operative Day 1 at 0700(T6). Central venous oxygen saturation measurements and mixed venous oxygen saturation using the PAC was also obtained at similar interval times as above. Low central venous oxygen saturation is defined as less than 70% while low mixed venous oxygen saturation was fixed as less than 65% for appropriate interventions to be instituted to improve oxygen delivery. Arterial blood gases will also be done at the scheduled interval to validate whether the presence of metabolic acidosis can be used to correlate with central or mixed venous oxygen saturation measurements.

MEASUREMENTS AND RESULTS: Demographic data that was recorded include age, sex, body weight, height, and body mass index, type of surgery, ejection fraction, time on cardiopulmonary bypass, Euroscore, haemoglobin and haematocrit levels.

At the scheduled interval, cardiac output measurements using the thermodilution method as well as the pulse contour analysis method using the Vigileo FloTrac system will be done. Mixed venous oxygen (SvO2) will be sampled simultaneously with the central venous oxygen saturation (ScvO2 ).

Demographic data will be summarized as mean ± SD where appropriate. Bland -Altman plot will be done to compare both methods for obtaining the cardiac output measurements. Linear regression analysis, Bland-Altman plot and Pearson test will be used to evaluate the correlation between SvO2 and ScvO2. A p-value of < 0.05 will be considered as significant.

EXCLUSION CRITERIA: Patients will be excluded if they are on Intra Aortic Balloon Pump (IABP), requiring emergency chest reopening, significant arrhythmia which causes an irregular arterial waveform and tricuspid regurgitation as ruled out during the pre operative echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing coronary bypass graft surgery and valvular heart disease.

Exclusion Criteria:

* Patients will be excluded if they are on Intra Aortic Balloon Pump (IABP), requiring emergency chest reopening, significant arrhythmia which causes an irregular arterial waveform and tricuspid regurgitation as ruled out during the pre operative echocardiogram.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Cardiac output and other haemodynamic indices | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Subrahmanyam Balan, MBBS, Study Chair — Hospital Sultanah Aminah Johor Bahru
Locations (1):
- Hospital Sultanah Aminah, Johor Bahru, Johor, Malaysia